CLINICAL TRIAL: NCT04323540
Title: Surgical Reconstructive Treatment of Peri-Implantitis With or Without Simultaneous Soft Tissue Augmentation: a Multi-center Randomized Controlled Trial
Brief Title: Treatment of Peri-implantitis With or Without Simultaneous Soft Tissue Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: George Eastman Dental Hospital, Italy (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Principal Investigator, Lucrezia Paternò Holtzman, Investigator, George Eastman Dental Hospital, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18117
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenograft+collagen membrane (Active Comparator): Reconstructive approach (Xenograft+collegen membrane)
  Interventions: Procedure: Peri-implantitis reconstructive surgery
- Xenograft+collagen membrane+autologous soft tissue graft (Experimental): Reconstructive approach (Xenograft+collegen membrane) plus soft tissue graft (autologous, harvested as FGG)
  Interventions: Procedure: Peri-implantitis reconstructive surgery

INTERVENTIONS:
Procedure: Peri-implantitis reconstructive surgery — For both arms (excluding the already included information): defect debridement, removal of debris using titanium curettes, titanium brushes on the implant surface, irrigation with saline, application of sterile cotton pellets with saline solution. Grafting with (experimental) xenograft and soft tissue, or xenograft alone (control). Suture.
  Specific to control group (active comparator): the peri-implant defect will be filled with xenograft, and a collagen membrane will be fitted and trimmed to the defect area.
  Specific to test/experimental group: same as above (for control). In addition a soft tissue graft will be harvested from the palate and sutured to the buccal flap. The entire flap will then be sutured to the lingual flap.

SUMMARY:
The study will aim to compare two modalities in the reconstructive treatment of peri-implantitis defects. More specifically, the control group will be a reconstructive approach (xenograft bone graft granules and collagen membrane, BioOss and BioGide, Geistlich, Wolhusen). The test group will be the same with the exception of an autologous sub-epithelial connective tissue palatal graft, sutured beneath the flap, which will be used in addition to grafting materials.

Outcomes will include CAL, PD, MR, defect resolution, PI, BoP, SUPP, patient-reported outcome measures including an aesthetic self-evaluation.

DETAILED DESCRIPTION:
The study will aim to compare two modalities in the reconstructive treatment of peri-implantitis defects.

More specifically, the control group will be a "pure" reconstructive approach (xenograft bone graft granules and reservable collagen membrane, BioOss and BioGide, Geistlich, Wolhusen). This is in accordance with gold standard practices of reconstructive therapy of peri-implant defects.

The test group will be treated with the same approach and materials, with the exception of an autologous sub-epithelial connective tissue palatal graft, sutured beneath the flap, which will be used in addition to the grafting materials. The graft will be harvested from the homolateral palate (molar region).

Outcomes will include CAL, clinical attachment level (primary outcome), PD or probing depth, MR or mucosal recession, defect resolution (composite outcome made up of simultaneous absence of PD>5 mm, BOP/SUP and bone level changes >0.5 mm, PI, BoP or bleeding upon probing, suppuration SUP on probing, SUP on palpation, patient-reported outcome measures including an aesthetic self-evaluation.

The measures will be recorded at baseline, 6-, 12-, 18- and 24 months. Radiographic bone levels will be compared with 2 week image at 12 and 24 months

ELIGIBILITY:
Inclusion Criteria:

* · Be able and willing to provide consent and sign the informed consent form.

  * Be able and willing to comply with study procedures and follow-up appointments required by the study protocol.
  * Age>18 years
  * Presence of at least one implant affected with peri-implantitis, defined as the following con-dition: at least one site presenting peri-implant probing depth (PPD) >6 mm and simultane-ous presence of profuse BoP/SUP and a radiographically documented change in bone level greater than initial bone remodeling. In the likely event that a baseline radiographic image is absent, the bone level will be compared to where it would likely have been at the time of implant insertion and a difference of >3 mm from that level will be considered.
  * Implants in function (i.e. loaded) for at least 1 year.
  * Screw- and cement-retained suprastructures for both fixed and removable prostheses.

Exclusion Criteria:

* Compromised systemic health which contraindicates the study procedures.
* Pregnant or nursing women.
* Cigarette smoking>5 per day
* Systemic conditions compromising healing (i.e. diabetes mellitus). Patients with diabe-tes mellitus types I or II will be asked to provide information regarding their most re-cent HbA1c values. Only patients with HbA1c<7% will be enrolled.
* Patients taking medications known to interfere with gingival or bone metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | change from baseline to: 6, 12, 18, 24 months
  linear distance (mm) from the implant platform to the bottom of the pocket

SECONDARY OUTCOMES:
Probing depth | 6, 12, 18, 24 months
  linear distance (mm) from the gingival margin to the bottom of the pocket
Disease resolution | 6, 12, 18, 24 months
  No PD greater than or equal to 5 mm and simultaneous absence of BOP/SUP and no more than 0.5 mm change between 2 weeks and 12 and 24 months on radiograph
Mucosal recession | 6, 12, 18, 24 months
  linear distance (mm) from the implant platform to the gingival margin
plaque index (minimum value 0, maximum 1) | 6, 12, 18, 24 months
  binary outcome: yes/ no detected running the probe into the peri-implant sulcus
profuse bleeding | 6, 12, 18, 24 months
  abundant bleeding evoked upon probing immediately after
BOP | 6, 12, 18, 24 months
  bleeding upon probing: bleeding evoked upon probing after 1 second
suppuration | 6, 12, 18, 24 months
  Binary: yes or no, detected upon probing or digital palpation
Gingival thickness | 6, 12, 18, 24 months
  Measured in a horizontal direction at 1 mm from the gingival margin
Patient-reported outcome measures | 6, 12, 18, 24 months
  pain-bleeding-aesthetic self-evaluation-swelling-discomfort
Radiographic bone levels | 2 weeks, 12 months, 24 months
  radiographic bone level changes between the 2 week and 12 and 24 month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cordaro, MD, PhD, Principal Investigator — G. Eastman Dental Hospital Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holtzman LP, Milinkovic I, Vuckovic M, Malpassi C, Cuppini M, Solderer A, Aleksic Z, Cordaro L. Effect of Connective Tissue Graft as an Adjunct to Guided Bone Regeneration in the Surgical Treatment of Peri-Implantitis: A Dual-Center Randomized Controlled Trial. Clin Oral Implants Res. 2026 Jan 31. doi: 10.1111/clr.70093. Online ahead of print. PMID 41618697